CLINICAL TRIAL: NCT03647813
Title: Effects of Photobiomodulation Therapy in Salivary Analysis of Chronic Renal Failure Patients Undergoing Hemodialysis: a Randomized Placebo-controlled Trial
Brief Title: Effects of Photobiomodulation in Salivary Analysis of Chronic Renal Failure Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vanessa
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Xerostomia; Chronic Renal Failure
MeSH Terms: conditions — Xerostomia; Kidney Failure, Chronic | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Only one researcher knew in which group the patients were allocated and performed all the treatments. A blinded researcher performed all the evaluations after the procedures. The patient was also blinded to the treatment as the laser was turned off, simulating the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation group (Active Comparator): Patients were submitted to three sessions of PBM (baseline, 7 and 14 days). PBMT was administered by a single professional using a continuous wave AsGaAl diode laser (Photon Lase III - DMC, São Paulo, Brazil) with a wavelength of 808 nm (infrared). Irradiation was performed in punctual contact mode (ʎ = 808 nm, 100 mW, 142 J/cm2 and 4 J per point). A total of 20 points were applied in each session/day being three extraoral points in the parotid region (right and left n=6), three points in buccal mucosa (right and left, n=6), two extraoral (right and left, n=4) and two intraoral (right and left, n=4) points in the submandibular and sublingual regions.
  Interventions: Radiation: Photobiomodulation
- Placebo group (Placebo Comparator): Patients were submitted to same protocol as the photobiomodulation group, but the laser was turned off.
  Interventions: Radiation: Placebo

INTERVENTIONS:
Radiation: Photobiomodulation — Patients received three irradiations of laser at ʎ = 808 nm, 100 mW, 142 J/cm2 and 4 J per point.
  Arms: Photobiomodulation group
Radiation: Placebo — The same laser protocol was followed but with the device switched off.
  Arms: Placebo group

SUMMARY:
End-stage renal disease patients undergoing hemodialysis can present alteration in flow, concentrations and composition of saliva affecting oral health. This randomized placebo-controlled trial aims to evaluate the effectiveness of photobiomodulation therapy (PBM) in salivary parameters in chronic renal failure (CRF) patients undergoing hemodialysis. Forty-four patients with CRF on hemodialysis self-responded two questionnaires for oral health and salivary gland function perception. Thereafter, patients were clinically evaluated for the diagnosis of hypofunction of salivary glands and were randomly allocated into two groups: PBM group (n = 21), which received three irradiations of laser at ʎ = 808 nm, 100 mW, 142 J/cm2 and 4 J per point; and a placebo group (n = 17) that consisted of laser protocol with the device switched off. Patients were first submitted to sialometry and after to PBM or placebo intervention at baseline, 7 and 14 days. Non-stimulated and stimulated saliva were collected for salivary volume investigation and biochemical analysis of total protein, calcium and urea concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Stable cardiopulmonary and neurological conditions;
* Hb> 10.9 g / dl and Hematocrit> 33;
* Absence of acute systemic infectious processes;
* Blood pressure <140 mmHg and PAd <90 mmHg in at least two measurements in two subsequent dialysis;
* No hypervolemia;
* Patients over 18 years-old;
* Signed a statement of informed consent.

Exclusion Criteria:

* Patients in intensive care unit;
* Hemodynamic instability, signs and symptoms of uremic syndrome related to the cardiovascular and neurological systems;
* Presence of acute systemic infectious processes;
* Presence of acute cardiovascular disease, systolic blood pressure > 141 mmHg and / or diastolic blood pressure > 91 mmHg;
* Significant anemia (Hb <11 g / dl and Hto <33%);
* Photosensitivity;
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Sialometry (measurement of the amount of produced saliva before and after treatment) | Baseline, 7 days and 14 days.
  Non-stimulated salivary collection was obtained with patient seated with heads slightly forward and a graduated collector tube positioned under the lower lip for 5 minutes to collect saliva. To obtain the stimulated saliva, patients stayed in the same position and chewed a piece of silicone of a standard size for 5 minutes. All the saliva produced was dispensed in another graduated tube. Salivary volumes were calculated using the difference in weight before and after collection provided a ratio with the volume in milliliters of expelled saliva. An analysis of salivary total proteins, urea and calcium levels were quantified in triplicates using colorimetric analysis with commercially available kits (Bioclin, Belo Horizonte, Minas Gerais,Brazil) and a spectrophotometer (Anthos 2020 - Asys - Austria) end point methods The absorbance for each marker was measured using the wavelength indicated by manufacture.